CLINICAL TRIAL: NCT01345409
Title: Acupuncture and Chiropractic Care for Chronic Pain in an Integrated Health Plan
Acronym: Relief
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Arizona (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01AT005896-01 (NIH)
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Pain
Keywords: Musculoskeletal pain; Chronic pain; Acupuncture; Chiropractic
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recent research examines many types of complementary and alternative (CAM) therapies. However, "real-world" use of CAM has been largely overlooked.

This project consists of four discrete sets of project activities (that largely follow one another chronologically).

Phase1 uses information from the EMR (patient electronic medical records) to identify unique clusters of patients with CMP (chronic musculoskeletal pain), their care within the health plan, and to examine how those in unique clusters may have different uses for A/C (acupuncture and chiropractic) services and/or differential outcomes associated with such care.

Phase 2 will conduct a survey of CMP patients from KPNW (Kaiser Permanente Northwest region) to establish a broad sample of patients and their use of out-of-plan CAM services.

Phase 3 will collect qualitative data (focus groups and individual interviews) from KP members, KP providers, and acupuncturists and chiropractors from the community to examine KP providers' decision to recommend A/C services, A/C services delivered to KP patients, and patients' decisions to pursue and retain CAM care. A secondary purpose is to have KP members with CMP review planned assessment instruments to improve understandability of the instruments. They will provide feedback on: relevancy, any notable omissions of domains important in patients' decision to use CAM services for pain treatment. They will also provide insight to broader health and quality of life outcomes associated with such CAM treatments.

Phase 4 is a prospective cohort study to evaluate health services/costs and broader clinical and functional outcomes associated with the receipt of A/C relative to carefully matched comparison participants receiving traditional CMP services.

DETAILED DESCRIPTION:
Substantial recent research examines the efficacy and biological basis of many types of complementary and alternative (CAM) therapies. However, "real-world" use of CAM has been largely overlooked, despite calls for CAM therapies to be studied in the manner in which they are practiced and urging high prioritization for research that includes clinical outcomes, cost-effectiveness, and the decision-making process for patients and providers. There is, therefore, heightened need for enriched understanding-particularly given CAM's growing popularity, which fortunately offers stores of new data for research. Recent studies suggests that Americans seek CAM treatments far more often for chronic musculoskeletal pain (CMP) than for any other condition. Among CAM treatments for CMP, acupuncture and chiropractic (A/C) care are among those with the highest acceptance by physician groups and the best evidence to support their use. Further, recent alarming increases in delivery of opioid treatment and surgical interventions for chronic pain-despite their high costs, potential adverse effects, and modest efficacy-suggests the need to evaluate the outcomes associated with promising non-pharmacological/non-surgical CAM treatments for CMP, which are often well accepted by patients and increasingly used in the community.

This study responds to the NCCAM program announcement PAR-08-045, "Outcomes, Cost-Effectiveness and the Decision Making Process to Use CAM."

Because this project consists of four discrete sets of project activities (that largely follow one another chronologically), the investigators plan to submit separate IRQs to cover each set of project activities as follows:

(Phase1) Retrospective study using information from the EMR to identify unique clusters of patients with CMP, their trajectories of care within the health plan, and to examine how those in unique clusters may have differing propensities for the use of A/C services and/or differential outcomes associated with such care. The IRQ for this study has been submitted (Phase 2) The administration of an out-of-plan CAM survey to determine from a broad sample of KP members their use of such services.

(Phase 3) The collection of qualitative data (focus groups and individual interviews) from KP members, KP providers, and acupuncturists and chiropractors from the community to examine KP providers decision to recommend A/C services, A/C services delivered to KP patients, and patients' decisions to pursue and retain CAM care. A secondary purpose is to have KP members with CMP review planned assessment instruments for phase 4 of the study to provide feedback on: relevancy, any notable omissions of domains important in patients' decision to use CAM services for pain treatment and broader health and quality of life outcomes associated with such CAM treatments, as well as to review understandability of the assessment instruments.

(Phase 4) A prospective cohort study to evaluate health services/costs and broader clinical and functional outcomes associated with the receipt of A/C relative to carefully matched comparison participants receiving traditional CMP services.

ELIGIBILITY:
Inclusion Criteria:

* KPNW health plan members
* 18 or older
* Evidence of CMP

Exclusion Criteria:

* Malignant cancer diagnosis
* Hospice or other end-of-life palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic musculoskeletal pain (CMP)
Sampling Method: Non-Probability Sample
Enrollment: 1242 (Actual)
Dates: Start 2010-12; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain severity & interference | Baseline, 1-, 3-, 6-months
  Two subscales -- the 4-item pain severity and the 7-item pain interference subscales -- from the short form of the Brief Pain Inventory (BPI-SF) will be used to assess pain and related disability.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn DeBar, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Penney LS, Ritenbaugh C, DeBar LL, Elder C, Deyo RA. Provider and patient perspectives on opioids and alternative treatments for managing chronic pain: a qualitative study. BMC Fam Pract. 2017 Mar 24;17(1):164. doi: 10.1186/s12875-016-0566-0. PMID 28403822
- [Derived] DeBar LL, Elder C, Ritenbaugh C, Aickin M, Deyo R, Meenan R, Dickerson J, Webster JA, Jo Yarborough B. Acupuncture and chiropractic care for chronic pain in an integrated health plan: a mixed methods study. BMC Complement Altern Med. 2011 Nov 25;11:118. doi: 10.1186/1472-6882-11-118. PMID 22118061